CLINICAL TRIAL: NCT04911777
Title: A Randomized, Double-Blind, Placebo-Controlled, Proof of Principle Study of Pentarlandir™ UPPTA for the Treatment of Patients With Early COVID-19
Brief Title: Proof of Principle Study to Evaluate the Safety, PK, Viral Shedding and Efficacy of Pentarlandir™ UPPTA for Patients With Early COVID-19
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: SyneuRx International (Taiwan) Corp (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: SNR08-Covid19
Record Dates: First submitted 2021-06-01; First posted 2021-06-03 (Actual); Last update posted 2021-12-17 (Actual); Status verified 2021-12

CONDITIONS: Coronavirus Disease 2019
Keywords: COVID-19; Pentarlandir™ UPPTA; UPPTA
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: In the first phase, 45 subjects will be randomized at 2:1 ratio to Pentarlandir™ UPPTA low dose or placebo. After interim analysis and evaluate by DSMB, 45 subjects will be randomized to 2:1 ratio to Pentarlandir™ UPPTA high dose or placebo in second phase. The final sample will be high-dose, low-dose, and placebo group at 1:1:1 ratio.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Pentarlandir™ UPPTA - High Dose (Experimental): High dose of Pentarlandir™ UPPTA, q8h (over 3 hours postprandially)
  Interventions: Drug: Pentarlandir™ UPPTA
- Pentarlandir™ UPPTA - Low Dose (Experimental): Low dose of Pentarlandir™ UPPTA and placebo, q8h (over 3 hours postprandially)
  Interventions: Drug: Pentarlandir™ UPPTA; Drug: Placebo
- Placebo (Placebo Comparator): Pacebo, q8h (over 3 hours postprandially)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pentarlandir™ UPPTA — Pentarlandir™ UPPTA is a white oral capsule (with 188 mg of UPPTA)
  Arms: Pentarlandir™ UPPTA - High Dose; Pentarlandir™ UPPTA - Low Dose
Drug: Placebo — The placebo of Pentarlandir™ UPPTA is a white oral capsule (without UPPTA)
  Arms: Pentarlandir™ UPPTA - Low Dose; Placebo

SUMMARY:
This is a clinical trial to evaluate the safety, PK, viral shedding and clinical effects of Pentarlandir™ UPPTA in patients with early COVID-19. Approximately 90 ambulatory subjects with mildly symptomatic early COVID-19, who have been diagnosed with COVID-19 within the prior 4 days will be enrolled.

DETAILED DESCRIPTION:
This is a clinical trial to evaluate the safety, PK, viral shedding and efficacy of PentarlandirTM UPPTA as a treatment for patients with early COVID-19. Approximately 90 ambulatory subjects with mildly symptomatic early COVID-19, who have been diagnosed with COVID-19 within the prior 48 hours, will be enrolled in the proof of principle study.

Upon signing informed consent and evaluating medical history, concomitant medications, oxygen saturation (SaO2) at room air and vital signs, a focused physical examination of the heart and lungs will be performed. Subjects will be randomized into High-Dose, Low-Dose, and Placebo group in a 1:1:1 ratio at the final sample, but the enrollment will be staggered. In the first phase, 45 study subjects will be randomized at 2:1 ratio to Pentarlandir™ UPPTA low dose or placebo. After all the forty-five (45) subjects have completed the Day 21 assessment or early terminated (14-day dosing and 7 days of followed-up), DSMB will review the safety from the cohort and provide concurrence with proceeding with the higher dose cohort. If DSMB deems that the study is safe to proceed, another 45 subjects will be randomized at 2:1 ratio to Pentarlandir™ UPPTA high dose or placebo in the second phase. Both staggered cohorts will have the same stopping rules.

During both phases of study, specimens for quantification of the viral genome, inflammatory markers, and safety laboratory tests will be collected. The IP will be dispensed to the study subjects and the subject will take the first dose of the study treatment at the clinic. Study subjects will be instructed (and provided) to use a device for ePRO for how to complete the patient-reported diary.

The subjects will take the IP orally. Subjects in the low-dose group will take from each bottle of the active drug and placebo every 8 hours (q8h); for the high-dose group, from each of the two bottles of active drug; and for the placebo group, from each of the two bottles of placebo for 14 days. The first treatment dose should be taken within 4 days of COVID-19 diagnosis. Physical examination, specimen collection, laboratory evaluations and urine pregnancy test, vital signs, pulse oxygen saturation and clinical symptom and status determination will be conducted.

Subjects who meet the eligibility criteria will be randomized. All subjects who fail to meet eligibility criteria are considered screen failures and are exited from the study without further evaluation.

Screening and Randomization (V1, Day 1):

After determining the eligibility, the study subjects will be randomized 2:1 to Pentarlandir™ UPPTA (either low or high dose) or placebo. The IP for treatment period will be dispensed to the study subjects and the subject will take the first dose of the study treatment at the study site. Study subjects will be instructed (and provided) how to complete the electronic patient reported outcome (ePRO) on a device.

Treatment Period (V2 - V14 (EOT), Day 2 - Day 14):

The subjects will continue to document the daily diary of ePRO. Total 13 visits are included in this period. Except 4 in-persons visits (V3, V7, V10, and V14), no in-person visit is expected during the study. Subjects will return to the clinical study sites to collect specimens for quantification of viral genome, inflammatory markers, pharmacokinetic and safety laboratory tests as well as record the SaO2, oral temperature, heart and respiratory rate, blood pressure, symptoms and concomitant medications, to document clinical status and adverse events (AEs), and IP accountability will be monitored. In addition, clinical symptom assessments and 7-category ordinal scale will be evaluated as well along with safety laboratory evaluations to determine whether the subject will continue to take the IP or stop the clinical trial. The subject will return the study treatment bottles at EOT visit.

Except for the in-person visits, subjects will be phone-called once every day between 8:00 AM and 7:00 PM on the visits to record concomitant medications and to document clinical status and 7-category ordinal scale as well as adverse events (AEs) to determine whether the subject will be taken of the IP and/or stop the clinical trial.

Weekly Follow-Up Period (V15 - V20, Day 15 - Day 56):

Between Day 15 to 28, subjects will perform the ePRO diary daily. In addition to ePRO, study subjects will be called every 7±2 days after EOT visit to document final outcome and AEs up to Day 56. AE/SAEs, hospital and ICU lengths of stays, and mortality in hospitalized subjects will be documented.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women 18 years of age or older.
2. Able and willing to provide informed consent.
3. Able and willing to sufficiently operate smart phones and study-provided monitoring devices per the Investigator.
4. Early COVID-19 diagnosis with mild severity defined as meeting all of the below:

   1. Confirmation of COVID-19 by a PCR-based diagnostic within 4 days of randomization.

      * COVID-19 with mild symptoms, defined as a score of 8 or higher on the clinical symptom score.
      * Clinical symptom score includes 9 items in fever or chills, myalgia, cough, headache, sore throat, new loss of test or smell, gastrointestinal symptoms (nausea, vomiting, diarrhea or abdominal pain), congestion or running nose, and fatigue (malaise) as assessed and recorded by the investigator.

      Note: The total score per patient ranges from 0 to 27 points. Each symptom is rated from 0 to 3. [0 = none, 1 = mild, 2 = moderate, and 3 = severe]
   2. No signs of a more serious lower airway disease per clinical exam, chest X-ray or chest CT.
   3. Resting RR ≤ 20, HR ≤ 90, oxygen saturation (pulse oximetry) ≥ 95% on room air.
5. For women of childbearing potential (women who are not permanently sterile [documented hysterectomy, bilateral tubal ligation, salpingectomy, or oophorectomy] or postmenopausal [12 months with no menses without an alternative medical cause]):

   1. Negative urine pregnancy test at screening.
   2. Willingness to practice a highly effective method of contraception that includes, but is not limited to, abstinence, sex only with persons of the same sex, monogamous relationship with a postmenopausal partner, monogamous relationship with vasectomize partner, vasectomy, licensed hormonal methods, intrauterine device, or consistent use of a barrier method (e.g., condom, diaphragm) with spermicide for 28 days after the last dose of study medication.
6. Ability and willingness to comply with all aspects of the study through the entire study period.

Exclusion Criteria:

1. Patient is either asymptomatic or with baseline severity of moderate, sever, or critical COVID-19.
2. Pregnant or lactating women.
3. Patients with shortness of breath at rest.
4. Findings on physical examination or available imaging studies suggesting rapid disease progression of COVID-19.
5. Signs or symptoms indicative of pneumonia or any other lower respiratory tract disorders, or clinically significant findings in available lung imaging studies suggestive of such disorders.
6. Need for immediate hospitalization, oxygen supplementation or mechanical ventilation.
7. Obstructive airway diseases, including chronic obstructive pulmonary disease (COPD) and asthma, or other respiratory disease that could exacerbate independent of COVID-19.
8. Use of remdesivir, chloroquine, hydroxychloroquine, convalescent plasma, other monoclonal antibody therapies, include REGEN-COV (casirivimab and imdevimab), bamlanivimab (plus etesevimab), dexamethasone, ivermectin, baricitinib, and other Janus kinase inhibitors, Bruton's tyrosine kinase inhibitors, tocilizumab (and other interleukin-6 inhibitors) and any other therapy with EUA or approval and other investigational agents for COVID-19.
9. Patients who are participating in other clinical trials.
10. History of conditions associated with immunocompromise, or treatments known to affect the immune system, including but not limited to oral or intravenous corticosteroids, alkylating drugs, antimetabolites, cytotoxic drugs, other chemotherapy, radiation, immune-modulating biologics, within 30 days of screening.
11. Barium enemas within the last 30 days.
12. Taking OTC or prescribed medicine which has compound as active ingredient.
13. Any unstable or uncontrolled medical illnesses such as neurological disorders, cardiovascular disorders, diabetes, hepatic or renal disorders that per the Investigator would intervene with the study conduct or study results interpretation.
14. Any other medical, psychiatric, or social condition or occupational or other responsibility that in the judgment of the Investigator would interfere with or serve as a contraindication to protocol adherence, assessment of safety, or a patient's ability to give informed consent or respond to the study procedures or questions during the personal visits or the video calls.
15. High-risk individuals are those who meet at least one of the following criteria:

    1. Aged ≥ 65 years
    2. Body mass index (BMI) > 30
    3. Pregnancy
    4. Chronic kidney disease
    5. Diabetes
    6. Immunosuppressive disease or immunosuppressive treatment
    7. Cardiovascular disease (including congenital heart disease) or hypertension
    8. Chronic lung diseases (for example, chronic obstructive pulmonary disease, asthma [moderate-to-severe], interstitial lung disease, cystic fibrosis and pulmonary hypertension)
    9. Sickle cell disease
    10. Neurodevelopmental disorders (for example, cerebral palsy) or other conditions that confer medical complexity (for example, genetic or metabolic syndromes and severe congenital anomalies)
    11. Having a medical-related technological dependence (for example, tracheostomy, gastrostomy, or positive pressure ventilation [not related to COVID-19]
    12. Exclusion is not limited to the medical conditions or factors listed above. The investigators have to consider the benefit-risk for an individual patient to determine other medical conditions or factors (for example, overweight, race or ethnicity) may also place individual patients at high risk for progression to severe COVID-19 and be excluded.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-08-24 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in viral genome up to Day 14 | Baseline and Day14

SECONDARY OUTCOMES:
Pharmacokinetics: Mean Concentration of Pentarlandir™ UPPTA on Days 3, 7, 10, 14. | Day 3, 7, 10, and 14
Change from baseline in daily COVID-19-related symptom severity score through Day 28 | Baseline to Day 28
  A set of common COVID-19-related symptoms (see patient diary template for electronic Patient Report Outcome (ePRO)) will be evaluated daily by the patient regardless of which symptoms he/she had at baseline, as new symptoms may appear following the baseline assessment. (A Likert symptom scale will be developed using the (The 24 items reported in the ePRO, with potentially each item being normalized to 0 to 3 and the total score ranging from ranged 0 to 72))
Number of days with substantial COVID-19-associated symptoms from start of study treatment (Day 1) based on self-assessment using daily symptom diary. | 28 days
  Substantial COVID-19-associated symptom days are defined as number of days when any symptoms score as moderate or sever in ePRO through Day 28
Number of days without COVID-19-associated symptoms in ePRO from Day 1-28 based on self- assessment using daily ePRO symptom diary. | 28 days
  Symptom-free days are defined as number of days when all the symptoms score as absent (or none) in ePRO through Day 28.
Number of days with limited COVID-19-associated symptoms in ePRO from Day 1-28 based on self- assessment using daily ePRO symptom diary. | 28 days
  Days with limited COVID-19-associated symptoms are defined as number of days when up to two symptoms score as mild or absent while the rest score as absent (or none) in ePRO through Day 28.
Number of days with progression (or worsening) of COVID-19-associated symptoms in ePRO through Day 28 compared to baseline. | Baseline to Day 28
  Progression or symptom worsening is defined as number of days when any symptoms scored as:
  1. moderate at baseline but score as severe on any day through Day28.
  2. mild at baseline but score as moderate or severe on any day through Day 28.
  3. absent at baseline but score as mild, moderate or worse on any day through Day 28.
Time to resolution, where resolution is defined as when a subject has scored absent (or none) on all COVID-19-associated symptoms for two consecutive days | 28 days
Patient-reported global impression in ePRO | 28 days
  Patient-reported global impression in ePRO includes the following "In general, would you say that your health is excellent, very good, fair, or poor?" (The scores will be ranged between 1-5; excellent to poor)
Change from baseline in the patient's health status on a 7-category ordinal scale at up to Day 14 | Baseline to Day 14
  A 7-category ordinal scale of patient health status ranges from 1) Death; 2) Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO); 3) Hospitalized, on non-invasive ventilation or high flow oxygen devices; 4) Hospitalized, requiring supplemental oxygen; 5) Hospitalized, not requiring supplemental oxygen; 6) Not hospitalized, limitation on activities; 7) Not hospitalized, no limitations on activities.
Change from baseline in pulse oxygen saturation up to Day 14 | Baseline to Day 14

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - Cullman Clinical Trials, Cullman, Alabama
  - Cactus Clinical Research, Inc., Gilbert, Arizona
  - Synergy Healthcare, Bradenton, Florida
  - Columbus Clinical Services, Miami, Florida
  - C'A Research, LLC, Miami, Florida
  - CTMD Research, Palm Springs, Florida
  - Eminat Research Group, Plantation, Florida
  - Elite Medical Research, Dallas, Texas
  - Diversified Medical Practices, Houston, Texas
  - Accurate Clinical Research, Houston, Texas
  - 1960 Family Practice, Houston, Texas
  - Ayinde Clinical Research, Irving, Texas